CLINICAL TRIAL: NCT01992393
Title: Targeted Self-Management for Epilepsy and Serious Mental Illness
Brief Title: Targeted Self-Management for Epilepsy and Serious Mental Illness (TIME)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Case Western Reserve University (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Principal Investigator, Martha Sajatovic, MD, Professor of Psychiatry, Case Western Reserve University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 11-12-17
Record Dates: First submitted 2013-11-14; First posted 2013-11-25 (Estimated); Results first posted 2022-09-28 (Actual); Last update posted 2022-09-28 (Actual); Status verified 2022-09

CONDITIONS: Epilepsy; Schizophrenia; Schizoaffective Disorder; Bipolar Disorder; Depression
Keywords: Epilepsy; Schizophrenia; Schizoaffective Disorder; Bipolar Disorder; Depression; Intervention; Treatment; Adherence
MeSH Terms: conditions — Epilepsy; Schizophrenia; Psychotic Disorders; Bipolar Disorder; Depression | interventions — Time

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- TIME (Experimental): This arm will receive the TIME intervention.
  Interventions: Behavioral: TIME
- Treatment as Usual (TAU) (No Intervention): This arm will receive treatment as usual.

INTERVENTIONS:
Behavioral: TIME — TIME consists of 12 group sessions in which patients with epilepsy and mental illness will be coached on techniques to help manage their conditions. There will also be four follow-up telephone sessions after the series of group sessions is completed. In addition, approximately half of the participants will participate in qualitative interviews.
  Arms: TIME

SUMMARY:
For this project we propose to refine the psychosocial intervention developed in phase one, based on input from key stakeholders, and to test the feasibility, acceptability and preliminary efficacy of the intervention. The proposed project addresses unmet public health needs for a historically hard-to-reach group of individuals with epilepsy and comorbid serious mental illnesses, and as the intervention is an adjunct to care that individuals with serious mental illness are already receiving, and uses staff already likely to be present in a care system, it is ideally suited for "real-world" implementation in people with epilepsy and serious mental illness (E-SMI).

The purpose of this study is to try and engage individuals with E-SMI to actively participate in illness self-management and treatment adherence that are crucial in minimizing the morbidity and mortality associated with both chronic mental disorders and chronic neurological conditions.

ELIGIBILITY:
Inclusion Criteria:

* Able to provide written consent
* Able to speak and understand English
* Age 18 and older
* Diagnosed with epilepsy
* Diagnosed with serious mental illness (DSM IV diagnosis of schizophrenia, schizoaffective disorder, bipolar disorder or chronic/recurrent depression confirmed with the Mini-International Neuropsychiatric Interview (MINI))
* Receive care at a community mental health center or other publicly funded community healthcare entity

Exclusion Criteria:

* Actively suicidal/homicidal individuals
* Individuals with dementia
* Unable to be rated on study rating scales
* Pregnant women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2013-09; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Martha Sajatovic, MD, Principal Investigator — Case Western Reserve University
Locations (1):
- University Hospitals Case Medical Center, Cleveland, Ohio, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: We used the electronic medical record from a large citywide healthcare system to preliminarily identify people with an epilepsy diagnosis and invited them to participate in the RCT.
Pre-assignment Details: 14 participants were excluded at Screening because they did not meet the inclusion criteria: 4 No SMI, 2 No epilepsy, 3 No show (unwilling to participate), 3 withdrew from study, 1 Single episode SMI,1 Pregnancy
Period: Baseline
Arm/Group | TIME | Treatment as Usual (TAU)
Started | 22 | 22
Completed | 21 | 22
Not Completed | 1 | 0
Period: Week 12 (3 Months)
Arm/Group | TIME | Treatment as Usual (TAU)
Started | 21 | 22
Completed | 19 | 18
Not Completed | 2 | 4
Period: Week 16 (4 Months)
Arm/Group | TIME | Treatment as Usual (TAU)
Started | 19 | 18
Completed | 19 | 16
Not Completed | 0 | 2

BASELINE CHARACTERISTICS:
Population: Individuals with epilepsy and comorbid mental illness.
Groups:
- Total: Total of all reporting groups
Arm/Group | TIME | Treatment as Usual (TAU) | Total
Number analyzed (Participants) | 22 | 22 | 44
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.00 (7.58) | 45.10 (14.18) | 48.25 (11.82)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 13 | 26
  Male | 9 | 9 | 18
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 1 | 3
  Not Hispanic or Latino | 20 | 21 | 41
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White/Caucasian | 8 | 8 | 16
  Black/ African American | 13 | 12 | 25
  Other | 1 | 2 | 3
Education Level [Count of Participants; unit: Participants]
  Less than a high school education | 7 | 4 | 11
  High school graduate, GED, or higher | 15 | 18 | 33
Employment Status [Count of Participants; unit: Participants]
  Unemployed | 7 | 4 | 11
  Unable to work | 9 | 10 | 19
  Other | 6 | 7 | 13
  Data Missing | 0 | 1 | 1
Marital Status [Count of Participants; unit: Participants]
  Married | 4 | 0 | 4
  Other | 18 | 22 | 40
Living Situation [Count of Participants; unit: Participants]
  Lives alone | 14 | 8 | 22
  Only adult in household | 2 | 1 | 3
  Lives with other adults | 5 | 11 | 16
  Homeless | 1 | 2 | 3
Income Level [Count of Participants; unit: Participants]
  Less than $25,000 | 21 | 21 | 42
  $25,000-$50,000 | 1 | 1 | 2
  More than $50,000 | 0 | 0 | 0
Seizure Type [Number; unit: seizures]
  Generalized | 16 | 14 | 30
  Partial | 5 | 6 | 11
  Unclassified | 1 | 2 | 3
  Other | 1 | 3 | 4
  Don't know/Not sure | 1 | 4 | 5
Mental Health Diagnosis [Count of Participants; unit: Participants]
  Depression | 7 | 6 | 13
  Bipolar Disorder | 7 | 9 | 16
  Schizophrenia | 8 | 7 | 15
Duration of Mental Health Disorder (in years) [Mean (Standard Deviation); unit: years] | 30.27 (17.35) | 22.85 (12.33) | 26.14 (15.76)
Duration of Epilepsy (in years) [Mean (Standard Deviation); unit: years] | 27.55 (16.48) | 25.43 (15.47) | 26.27 (15.74)
Charlson Comorbidity Index (CCI) [Mean (Standard Deviation); unit: scores on a scale] — Self-reported Charlson Comorbidity Index (CCI) is comprised of the presence of 10 medical conditions including respiratory diseases, rheumatological diseases, cancer, diabetes, digestive problems, heart trouble, HIV/ AIDS, kidney disease, liver disease, & stroke. Total Score is the sum of all 10-items, each item checked gets 1 point, except heart disease & kidney disease which get 2 points each, liver disease gets 3 points, and cancer & HIV/AIDS which get 6 points each. The CCI summary score range from 0-24. A higher score is associated with increased risk of mortality.
  scores on a scale | 3.14 (2.47) | 1.86 (2.29) | 2.45 (2.44)
Rapid Estimate of Adult Literacy in Medicine-Revised (REALM-R) [Mean (Standard Deviation); unit: scores on a scale] — The Rapid Estimate of Adult Literacy in Medicine-Revised (REALM-R) is an 11 item measure that identifies patients that are at high risk for having limited health literacy and identifies the grade level of the patient if they read below the ninth grade level.
  Each correctly pronounced word gets 1 point. The REALM-R Total Score is the sum of correct word pronunciations. With a total score ranging from 0 to 11. A score of 6 or less indicates risk for poor health literacy.
  scores on a scale | 5.18 (2.77) | 6.29 (2.57) | 5.77 (2.69)

OUTCOME MEASURES:

1. Primary Outcome: Change in Montgomery Asberg Depression Rating Scale (MADRS)
Description: The MADRS measures symptoms of depression. Total scores on MADRS range from 0-60, with higher scores indicating more severe depression.
Time Frame: Baseline to Week 16
Population: Individuals with epilepsy and comorbid mental illness.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | TIME | Treatment as Usual (TAU)
Number analyzed (Participants) | 22 | 22
score on a scale
  Baseline | 16.75 (10.28) | 22.94 (11.81)
  Week 16 | 11.21 (9.36) | 21.81 (10.50)
Statistical Analysis 1: Comparison: TIME vs Treatment as Usual (TAU); Test type: Other; p = 0.036, GEE

2. Secondary Outcome: World Health Organization Disability Assessment (WHODAS II)
Description: The World Health Organization Disability Assessment Schedule (WHODAS 2.0) assess functioning and disabilities in activities of daily living, including mobility, self-care, and life activities.
  Sum Scores from 32-180 with higher scores indicating greater degree of disability.
Time Frame: Baseline, 12 Week, 16 Week
Population: Individuals with epilepsy and comorbid mental illness with available data.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | TIME | Treatment as Usual (TAU)
Number analyzed (Participants) | 21 | 19
score on a scale
  Baseline | 80.86 (18.76) | 82.83 (23.39)
  12 week: number analyzed (Participants) | 17 | 15
  12 week | 67.68 (13.29) | 79.87 (24.44)
  16 week: number analyzed (Participants) | 18 | 14
  16 week | 73.39 (24.94) | 81.50 (21.34)
Statistical Analysis 1: Comparison: TIME vs Treatment as Usual (TAU); A two-sided two sample t-test comparing difference of values from baseline and 12 week between TIME and TAU; Test type: Other; p = 0.042, t-test, 2 sided
Statistical Analysis 2: Comparison: TIME vs Treatment as Usual (TAU); A two-sided two sample t-test comparing difference of values from baseline and 16 week between TIME and TAU; Test type: Other; p = 0.204, t-test, 2 sided

3. Secondary Outcome: Quality of Life Questionnaire (QOLIE-10)
Description: The QOLIE-10-P is a self-administered questionnaire and comprises 7 components including seizure worry, overall quality of life, emotional well-being, energy-fatigue, cognitive functioning, medication effect, and social function. The sum score is used in the analysis. Scores from 1-5 with lower scores indicating the least amount of problems
Time Frame: Baseline, 12 Week, 16 Week
Population: Individuals with epilepsy and comorbid mental illness with available data.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | TIME | Treatment as Usual (TAU)
Number analyzed (Participants) | 22 | 21
units on a scale
  Baseline | 2.85 (0.82) | 3.34 (0.25)
  12 Week: number analyzed (Participants) | 18 | 17
  12 Week | 2.38 (0.60) | 3.03 (0.79)
  16 Week: number analyzed (Participants) | 18 | 15
  16 Week | 2.56 (0.89) | 2.84 (0.73)
Statistical Analysis 1: Comparison: TIME vs Treatment as Usual (TAU); A two-sided two sample t-test comparing difference of values from baseline and 12 week between TIME and TAU; Test type: Other; p = 0.129, t-test, 2 sided
Statistical Analysis 2: Comparison: TIME vs Treatment as Usual (TAU); A two-sided two sample t-test comparing difference of values from baseline and 16 week between TIME and TAU; Test type: Other; p = 0.978, t-test, 2 sided

4. Secondary Outcome: Patient Health Questionnaire (PHQ-9)
Description: Scores from 0-27 with higher scores indicating more severe depressive symptoms.
Time Frame: Baseline, 12 Week, 16 Week
Population: Individuals with epilepsy and comorbid mental illness with available data.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | TIME | Treatment as Usual (TAU)
Number analyzed (Participants) | 20 | 21
score on a scale
  Baseline | 9.70 (5.55) | 11.76 (5.72)
  12 Week: number analyzed (Participants) | 17 | 16
  12 Week | 9.24 (4.97) | 13.19 (5.67)
  16 Week: number analyzed (Participants) | 16 | 15
  16 Week | 6.38 (4.44) | 12.87 (6.63)
Statistical Analysis 1: Comparison: TIME vs Treatment as Usual (TAU); A two-sided two sample t-test comparing difference of values from baseline and 12 week between TIME and TAU; Test type: Other; p = 0.128, t-test, 2 sided
Statistical Analysis 2: Comparison: TIME vs Treatment as Usual (TAU); A two-sided two sample t-test comparing difference of values from baseline and 16 week between TIME and TAU; Test type: Other; p = 0.015, t-test, 2 sided

5. Secondary Outcome: Pittsburgh Sleep Quality Index (PSQI)
Description: The PSQI contains 19 self-rated questions that are combined to form seven "component" scores each with a range of 0-3 points. In all cases, a score of "0" indicates no difficulty, while a score of "3" indicates severe difficulty. The seven component scores are then added to yield one "global" score, with a range of 0-21, "0" indicating no difficulty and "21" indicating severe difficulties in all areas (with higher scores indicating worse sleep quality).
Time Frame: Baseline, 12 Week, 16 Week
Population: Individuals with epilepsy and comorbid mental illness with available data.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | TIME | Treatment as Usual (TAU)
Number analyzed (Participants) | 20 | 20
score on a scale
  Baseline | 10.55 (4.49) | 12.95 (4.38)
  12 Week: number analyzed (Participants) | 16 | 14
  12 Week | 8.88 (3.30) | 12.21 (2.64)
  16 Week: number analyzed (Participants) | 13 | 11
  16 Week | 6.85 (3.80) | 11.45 (3.27)
Statistical Analysis 1: Comparison: TIME vs Treatment as Usual (TAU); A two-sided two sample t-test comparing difference of values from baseline and 12 week between TIME and TAU; Test type: Other; p = 0.759, t-test, 2 sided
Statistical Analysis 2: Comparison: TIME vs Treatment as Usual (TAU); A two-sided two sample t-test comparing difference of values from baseline and 16 week between TIME and TAU; Test type: Other; p = 0.471, t-test, 2 sided

6. Secondary Outcome: Brief Psychiatric Rating Scale (BPRS)
Description: The BPRS is a tool clinicians or researchers use to measure psychiatric symptoms such as anxiety, depression, and psychoses. The BPRS assesses the level of 18 symptom constructs such as hostility, suspiciousness, hallucination, and grandiosity. It is particularly useful in gauging the efficacy of treatment in patients who have moderate to severe psychoses. The total Score is the sum of all 18-items. Score ranges from 18-126 with higher scores indicating more psychiatric symptoms.
Time Frame: Baseline, 12 Week, 16 Week
Population: Individuals with epilepsy and comorbid mental illness with available data.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | TIME | Treatment as Usual (TAU)
Number analyzed (Participants) | 21 | 20
score on a scale
  Baseline | 36.90 (11.78) | 37.85 (10.39)
  12 Week: number analyzed (Participants) | 18 | 16
  12 Week | 33.89 (9.67) | 35.81 (11.24)
  16 Week: number analyzed (Participants) | 17 | 15
  16 Week | 29.59 (11.36) | 35.73 (9.63)
Statistical Analysis 1: Comparison: TIME vs Treatment as Usual (TAU); A two-sided two sample t-test comparing difference of values from baseline and 12 week between TIME and TAU; Test type: Other; p = 0.775, t-test, 2 sided
Statistical Analysis 2: Comparison: TIME vs Treatment as Usual (TAU); A two-sided two sample t-test comparing difference of values from baseline and 16 week between TIME and TAU; Test type: Other; p = 0.433, t-test, 2 sided

7. Secondary Outcome: Global Assessment of Functioning (GAF)
Description: The GAF assesses psychological, social and occupational functioning on a hypothetical continuum of mental health illness. Scores range from 0-100 with higher scores indicating higher global functioning.
Time Frame: Baseline, 12 Week, 16 Week
Population: Individuals with epilepsy and comorbid mental illness with available data.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | TIME | Treatment as Usual (TAU)
Number analyzed (Participants) | 22 | 21
score on a scale
  Baseline | 59.23 (17.06) | 54.57 (13.66)
  12 Week: number analyzed (Participants) | 18 | 17
  12 Week | 62.83 (15.98) | 59.00 (16.78)
  16 Week: number analyzed (Participants) | 18 | 16
  16 Week | 69.50 (18.27) | 59.94 (18.38)
Statistical Analysis 1: Comparison: TIME vs Treatment as Usual (TAU); A two-sided two sample t-test comparing difference of values from baseline and 12 week between TIME and TAU; Test type: Other; p = 0.936, t-test, 2 sided
Statistical Analysis 2: Comparison: TIME vs Treatment as Usual (TAU); A two-sided two sample t-test comparing difference of values from baseline and 16 week between TIME and TAU; Test type: Other; p = 0.600, t-test, 2 sided

8. Secondary Outcome: Seizure Frequency - Past 30 Days
Description: Self reported seizure frequency in the past 30 days
Time Frame: Baseline, 12 Week, 16 Week
Population: Individuals with epilepsy and comorbid mental illness with available data.
Measure: Mean (Standard Deviation); unit: number of seizures
Arm/Group | TIME | Treatment as Usual (TAU)
Number analyzed (Participants) | 18 | 16
number of seizures
  Baseline: number analyzed (Participants) | 18 | 14
  Baseline | 3.67 (14.08) | 8.79 (32.01)
  12 Week: number analyzed (Participants) | 18 | 15
  12 Week | 1.50 (2.68) | 18.40 (42.36)
  16 Week: number analyzed (Participants) | 17 | 16
  16 Week | 1.00 (1.97) | 6.44 (15.21)
Statistical Analysis 1: Comparison: TIME vs Treatment as Usual (TAU); A two-sided two sample t-test comparing difference of values from baseline and 12 week between TIME and TAU; Test type: Other; p = 0.560, t-test, 2 sided
Statistical Analysis 2: Comparison: TIME vs Treatment as Usual (TAU); A two-sided two sample t-test comparing difference of values from baseline and 12 week between TIME and TAU; Test type: Other; p = 0.305, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: All adverse events will be reviewed by study Principal Investigators on an ongoing basis during the study period of 4 months.
Arm/Group | TIME | Treatment as Usual (TAU)
All-Cause Mortality (participants affected / at risk) | 0/22 | 0/22
Serious Adverse Events (participants affected / at risk) | 12/22 | 1/22
Other Adverse Events (participants affected / at risk) | 2/22 | 0/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TIME (N=22) | Treatment as Usual (TAU) (N=22)
Suicide attempt (Nervous system disorders) | 0 (0) | 1 (1)
Seizures (Nervous system disorders) | 4 (4) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 0 (0) — Low blood pressure
Heart condition (Cardiac disorders) | 3 (3) | 0 (0)
Blood Sugar (Blood and lymphatic system disorders) | 1 (1) | 0 (0) — elevated blood sugar
Irritable Bowel Syndrome (Gastrointestinal disorders) | 1 (1) | 0 (0)
Mini Stroke (Cardiac disorders) | 1 (1) | 0 (0)
Limb amputation (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) — leg amputated due to complications of vascular surgery.
Circulatory Surgery (Surgical and medical procedures) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TIME (N=22) | Treatment as Usual (TAU) (N=22)
Surgeries (Surgical and medical procedures) | 1 (1) | 0 (0) — Outpatient surgery for the arm.
Foot issue (General disorders) | 1 (1) | 0 (0) — Swollen and painful foot, treated and released.

LIMITATIONS AND CAVEATS:
Limitations included small sample size & a single-site setting which may not be representative of people with E-MI. Those who agree to participate in a clinical trial may be more help-seeking than individuals with E-MI more broadly. We excluded individuals too psychiatrically ill to participate in groups. Additionally, raters were not blind to randomization assignment, we did not collect information on psychotropic medication changes or adherence, & epilepsy diagnosis was not verified with EEG.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No